CLINICAL TRIAL: NCT00117442
Title: An Open-Label, Randomised Study of Multi-Cycle, Dose Intensive Carboplatin/Paclitaxel With Pegfilgrastim Supported by Haematopoietic Progenitor Cell Re-Infusion in Whole Blood
Brief Title: A Study of Carboplatin/Paclitaxel With Pegfilgrastim Supported by Haematopoietic Progenitor Cell Re-Infusion in Whole Blood
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20010191
Record Dates: First submitted 2005-06-30; First posted 2005-07-07 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Breast Cancer; Lung Cancer; Ovarian Cancer
Keywords: solid tumour; unknown primary tumour; carboplatin; paclitaxel
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Ovarian Neoplasms | interventions — Carboplatin; Paclitaxel; pegfilgrastim

ARMS (4):
- Pegfilgrastim 18 mg (Experimental): Pegfilgrastim 18 mg given once for mobilization
  Interventions: Drug: carboplatin; Drug: paclitaxel; Drug: pegfilgrastim
- Filgrastim (Active Comparator): Filgrastim given daily for mobilization
  Interventions: Drug: carboplatin; Drug: paclitaxel
- Pegfilgrastim 12 mg (Experimental): Pegfilgrastim 12 mg given once for mobilization
  Interventions: Drug: carboplatin; Drug: paclitaxel; Drug: pegfilgrastim
- Pegfilgrastim 6 mg (Experimental): Pegfilgrastim 6 mg given once for mobilization
  Interventions: Drug: carboplatin; Drug: paclitaxel; Drug: pegfilgrastim

INTERVENTIONS:
Drug: carboplatin — Chemotherapy
Drug: paclitaxel — chemotherapy
Drug: pegfilgrastim — Growth factor for mobilization
  Arms: Pegfilgrastim 12 mg; Pegfilgrastim 18 mg; Pegfilgrastim 6 mg

SUMMARY:
The purpose of this study is to provide dose-finding information regarding the efficacy and kinetics of peripheral blood progenitor cell (PBPC) mobilisation by pegfilgrastim and to determine if carboplatin/paclitaxel can be delivered at a reduced cycle interval when supported by pegfilgrastim-mobilised PBPCs in whole blood.

ELIGIBILITY:
Inclusion Criteria: - Pathologically confirmed diagnosis of malignancy (solid tumour) suitable for treatment with intensified carboplatin and paclitaxel - Previously untreated with chemotherapy or radiotherapy - ECOG performance status 0 to 2 inclusive - Life expectancy greater than or equal to 12 weeks - ANC greater than or equal to 2.0 x 10^9/L, platelets greater than 100 x 10^9/L - Glomerular filtration rate greater than 60 mL/min Exclusion Criteria: - Active infection requiring treatment with systemic (IV or oral) anti-infectives (antibiotic, antifungal, antiviral) within 72 hours of randomisation - Known to be HIV positive - Any premalignant myeloid condition or any malignancy with myeloid characteristics (e.g., myelodysplastic syndromes, acute or chronic myelogenous leukaemia) - Prior malignancy within the last 5 years, with the exception of surgically cured basal/squamous skin cell carcinoma, and/or carcinoma of the cervix in-situ - History of impaired cardiac status [e.g., severe heart disease (NYHA greater than 2), cardiomyopathy, or congestive heart failure] - Bone marrow involvement of disease - Major surgery within 2 weeks before randomisation - Known sensitivity to E. coli derived drug products (e.g., filgrastim) - Previous exposure to pegfilgrastim

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2002-08; Primary Completion 2004-08 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
PBPC mobilization profiles and success rate of achieving planned chemotherapy administration on time. | Cycle 0, and through 4 cycles

SECONDARY OUTCOMES:
PBPC kinetics and response to chemotherapy treatment | Cycles 1-4

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Willis F, Theti D, Dean S, Bacon P, Baker N, Pettengell R. Pegfilgrastim successfully mobilizes megakaryocyte progenitors into the peripheral blood in subjects with solid tumours. Bone Marrow Transplant. 2008 Aug;42(3):167-73. doi: 10.1038/bmt.2008.147. Epub 2008 May 26. PMID 18500375
- [Result] Willis F, Woll P, Theti D, Jamali H, Bacon P, Baker N, Pettengell R. Pegfilgrastim for peripheral CD34+ mobilization in patients with solid tumours. Bone Marrow Transplant. 2009 Jun;43(12):927-34. doi: 10.1038/bmt.2008.411. Epub 2009 Jan 26. PMID 19169289
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_11_GCSFSD01_20010191.pdf
- See also: FDA-approved Drug Labeling — http://www.neulasta.com/
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf